CLINICAL TRIAL: NCT07408115
Title: Effect of the Dietary Supplement Bonafide-HF3.0 on Women Who Experience Vasomotor Symptoms: An Open Label Experience Trial
Brief Title: Herbal Dietary Supplementation on Vasomotor Symptoms in Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bonafide Health (Industry)
Responsible Party: Principal Investigator, Trisha VanDusseldorp, Dr. Trisha VanDusseldorp, Principle Investigator, Bonafide Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-HF-BT-0003
Record Dates: First submitted 2025-11-24; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hot Flashes; Hot Flash; Hot Flushes, Menopause, Postmenopause; Hot Flushes and/or Sweats; Hot Flushes; Night Sweats; Vasomotor Symptoms; Vasomotor Symptoms (VMS); Vasomotor Symptoms Associated With Menopause
Keywords: Postmenopausal; Post menopause; Vasomotor Symptoms; Night sweats; Hot Flashes; Hot Flushes; Non-hormonal Treatment; Supplement
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active: JDS-HF3.0 Active Group (Experimental): All participants supplementing with JDS-HF3.0
  Interventions: Dietary Supplement: JDS-HF3.0

INTERVENTIONS:
Dietary Supplement: JDS-HF3.0 — Active Supplement JDS-HF3.0

SUMMARY:
The goal of this study is to evaluate the efficacy of a neurokinin 1,3 antagonist on improving vasomotor symptoms (VMS) and overall menopause symptoms in women between the ages of 40-70. The primary research question is whether taking the study product daily for 4 weeks with an optional 8 week extension, significantly reduces the severity and frequency of menopause-related symptoms.

DETAILED DESCRIPTION:
About 200 women across the U.S. will take part in this open label trial. All participants will take the study product and will be instructed to consume two tablets each morning for 4 weeks. Participants will be offered the option to enroll in an 8 week extension after the 4 week supplementation period. During this extension, participants will be asked to continue supplementing with the study product at the same dosing regimen. If a participant opts out of the extension, the total time the participant will be in the study is 5 weeks, including baseline data collection. If a participant opts into the 8 week extension, the total time the participant will be in the study is 12 weeks.

This is a remotely-delivered trial with no in-person assessments. Participants will take part in four virtual check-ins, including a pre-screening visit, a screening visit, a baseline visit, and a initial end of study visit. If a participant opts into the 8 week extension, there will be two additional virtual visits that are each conducted 4 weeks apart, including a end-of-extension visit. Throughout the study, participants will be asked to complete daily diaries and weekly and monthly questionnaires to report on their symptoms and how they are feeling. Questions included in these assessments ask about hot flashes, night sweats, physical comfort, and overall well-being. The study is led by a research team based in Harrison, NY, USA.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women who are 40 to 70 years of age (inclusive).
2. Have a body mass index (BMI) between 18.5 to 34.9 kg/m2 (inclusive).
3. Have self-reported menopausal symptoms for the past 6 months.
4. Have self-reported ≥5 moderate to severe hot flashes per day, on average for 7 days.
5. In good general health (no active or uncontrolled diseases or conditions) and able to consume the study product.
6. Agree to refrain from treatments listed in the defined timeframe.
7. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant, or planning to become pregnant during the study.
2. Use of any treatment for menopausal symptoms or other concomitant treatments listed.
3. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
4. Received a vaccine for COVID-19 in the two weeks prior to screening or during the study period, current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually three months from the onset of COVID-19 with symptoms that last for at least two months and cannot be explained by an alternative diagnosis).
5. Have a positive medical history of heart disease, renal disease, hepatic impairment, or active systemic infection (i.e., Lyme disease, TB, HIV).
6. History of cancer (except localized skin cancer without metastases) within two years prior to screening.
7. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study or influence the results or the potential subject's ability to participate in the study.
8. History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (i.e., Crohn's disease, short bowel, acute or chronic pancreatitis, gastric bypass procedures, or pancreatic insufficiency).
9. Active vaginal infections/abnormalities (e.g., active urinary tract infection (UTI), genital hemorrhage of unknown origin, pelvic inflammatory disease (PID)). Note: screened participants with infections would be eligible to participate two weeks after completing their treatment (wash-out period).
10. Participant has an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
11. Major surgery in three months prior to screening or planned major surgery during the study.
12. History of alcohol or substance abuse in the last 5 years.
13. Use of any vaginal medications, cooling devices, cooling mattresses, cooling sprays, or patches purposed for hot flash control (i.e., V-qool patch, estrogen cream, etc.) one week before and during study. Note: Screened participants that are willing to undergo a washout of at least two weeks or possibly longer and abstain from using above products during the duration of their participation will be enrolled.
14. Previous participation in a Bonafide Health run clinical trial on Hot Flashes using Bonafide HF-3.0.
15. Participation in another clinical or research trial.
16. Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.
17. Currently incarcerated prisoners.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender Female
Enrollment: 112 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Hot Flash Symptoms assessed by the number and severity of hot flashes and times awakened at night due to night sweats collected via participant diary tracking electronically. | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  Study diary will be completed by participants daily from Day -7 to -1 to establish a pre-dose baseline and then from Day 1 to Day 28 ± for the initial study duration. If a participant participates in the optional extension, they will be asked to continue completing the diaries for an additional 56 ± 3 days, for a total of 84 ± 3 days. The information recorded will be the number and severity of hot flashes that occurred, the number of night sweats and severity, any changes in concomitant medication/dietary supplement information, and any changes in health (Day 1 to 84 ± 3). Efficacy outcomes include daily diary results (number and severity of hot flashes and number of times awakened at night due to night sweats)
Change from Baseline on Hot Flash Symptoms assessed via Hot Flash Related Daily Interference Scale (HFRDIS) scores. | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  The HFRDIS measures the impact of hot flashes on overall quality of life and nine specific activities (work, social activities, sleep, mood, leisure activities, concentration, enjoyment of life, sexuality, and relations with others).The rating scale ranges from 0-10, with 0 being does not interfere, and 10 being completely interferes. A higher score indicates a worse outcome.
Change from Baseline on Hot Flash Symptoms assessed via the Visual Analog Scale Vasomotor Symptoms Questionnaire (VAS). | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  The Visual Analog Scale (VAS) has symptoms recorded on a 10-cm line that represents a continuum between the two ends of a scale -"not bothered" on the left end (0cm) of the scale and "extremely bothered" on the right end (10 cm) of the scale. Subjects mark one point on that continuum, and researchers measure the distance from that point to one of the ends of the scale. Response options range from 0-100, with a higher score reflecting the worse outcome.
Change from Baseline on Overall Menopausal Symptoms assessed via the Greene Climacteric Scale (CGS). | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  The GCS was a scale created to be a brief and standardized method to measure climacteric symptoms or complaints. Each of the 21 items is scored between 0-3, with 0 being not at all bothered and 3 being extremely bothered. There are three sub-scales that are measured, which include vasomotor, physical and psychological symptoms. Responses with a higher score reflect a worse outcome.
Change from Baseline on Overall Menopausal Symptoms assessed via the Menopause Rating Scale (MRS). | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  The MRS is a self-administered scale that scores eleven items on a 5-point scale, with 0 being no complaints and 4 being very severe symptoms. Each question is rated on a 5-point scale, with the higher number correlating with the more severe symptoms and worse outcome.
Change from Baseline on Overall Menopausal Symptoms assessed via the Visual Analog Scale Vasomotor Symptoms Questionnaire (VAS). | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  The Visual Analog Scale (VAS) has symptoms recorded on a 10-cm line that represents a continuum between the two ends of a scale -"not bothered" on the left end (0cm) of the scale and "extremely bothered" on the right end (10 cm) of the scale. Subjects mark one point on that continuum, and researchers measure the distance from that point to one of the ends of the scale. Response options range from 0-100, with a higher score reflecting the worse outcome.

SECONDARY OUTCOMES:
Change from Baseline of Sleep Quality assessed via the Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form (PROMIS SD SF). | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  The Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form (PROMIS SD SF) assesses self-reported perceptions of sleep, including difficulties and concerns with getting to sleep or staying asleep, satisfaction of sleep, and overall sleep quality. This form does not focus on symptoms of specific sleep disorders; it is universal rather than disease-specific. It assesses sleep disturbance over the past seven days
Change from Baseline of Quality of Life assessed via the menopause-specific quality of life (MENQOL) | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  The MENQOL is a quality-of-life questionnaire that is specific to postmenopausal women.There are 29 questions that ask questions pertaining to symptoms or problems that are directly related to menopause. Each question being scored from 0 to 6, 0 being not at all bothered and 6 being extremely bothered, with 6 being the worse outcome.
Change from Baseline on Joint pain and discomfort assessed via the Joint Questionnaire | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  Change from baseline in scores in the Joint Questionnaire. The Joint Questionnaire is a modified version of the validated Musculoskeletal Questionnaire to include more relevant and joint pain/discomfort specific questions. The questionnaire contains eight questions focused on joint and/or muscular pain, discomfort, and or soreness in the past two weeks. Questions include multiple-choice answers based on severity and frequency.

OTHER OUTCOMES:
Safety and Tolerability assessed via participant electronic diaries | From enrollment to initial end of study at 8 weeks and/or end of study at optional 12 weeks
  Safety and adverse events (e.g., GI distress, headaches) will be collected from participant electronic diaries or in the event there is an adverse event that a participant contacts the study team this will be documented directly by the study team. Each virtual visit will also include a safety/adverse event check in with a study team member.

CONTACTS AND LOCATIONS:
Locations (1):
- Bonafide Health, Harrison, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be privately owned.

REFERENCES:
- [Background] Curet LB. Determination of gestational age. Wis Med J. 1979 Nov;78(11):43-4. No abstract available. PMID 516787
- [Background] O'Boyle KM, Waddington JL. Structural determinants of selective affinity for brain D-1 dopamine receptors within a series of 1-phenyl-1H-3-benzazepine analogues of SK&F 38393 and SCH 23390. Eur J Pharmacol. 1985 Sep 24;115(2-3):291-5. doi: 10.1016/0014-2999(85)90702-2. PMID 2866103
- [Background] Fazekas AT, Homoki J, Pal SB, Teller W, Pfeiffer EF. Effect of age and sex on cortisol concentrations of peripheral tissues and adrenals in white guinea pigs. Acta Endocrinol Suppl (Copenh). 1973;173:32. doi: 10.1530/acta.0.072s032. No abstract available. PMID 4542113
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Hilditch JR, Lewis J, Peter A, van Maris B, Ross A, Franssen E, Guyatt GH, Norton PG, Dunn E. A menopause-specific quality of life questionnaire: development and psychometric properties. Maturitas. 1996 Jul;24(3):161-75. doi: 10.1016/s0378-5122(96)82006-8. PMID 8844630
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Greene JG. Constructing a standard climacteric scale. Maturitas. 1998 May 20;29(1):25-31. doi: 10.1016/s0378-5122(98)00025-5. PMID 9643514
- [Background] Carpenter JS. The Hot Flash Related Daily Interference Scale: a tool for assessing the impact of hot flashes on quality of life following breast cancer. J Pain Symptom Manage. 2001 Dec;22(6):979-89. doi: 10.1016/s0885-3924(01)00353-0. PMID 11738160
- [Background] Scoglio S, Benedetti S, Canino C, Santagni S, Rattighieri E, Chierchia E, Canestrari F, Genazzani AD. Effect of a 2-month treatment with Klamin, a Klamath algae extract, on the general well-being, antioxidant profile and oxidative status of postmenopausal women. Gynecol Endocrinol. 2009 Apr;25(4):235-40. doi: 10.1080/09513590802632506. PMID 19408172
- [Background] https://doi.org/10.1177/20533691231172565
- [Background] Greene JG. Constructing a standard climacteric scale. Maturitas. 2008 Sep-Oct;61(1-2):78-84. doi: 10.1016/j.maturitas.2008.09.011. PMID 19434881
- [Background] Bannu SM, Lomada D, Gulla S, Chandrasekhar T, Reddanna P, Reddy MC. Potential Therapeutic Applications of C-Phycocyanin. Curr Drug Metab. 2019;20(12):967-976. doi: 10.2174/1389200220666191127110857. PMID 31775595
- [Background] Ataei-Almanghadim K, Farshbaf-Khalili A, Ostadrahimi AR, Shaseb E, Mirghafourvand M. The effect of oral capsule of curcumin and vitamin E on the hot flashes and anxiety in postmenopausal women: A triple blind randomised controlled trial. Complement Ther Med. 2020 Jan;48:102267. doi: 10.1016/j.ctim.2019.102267. Epub 2019 Nov 26. PMID 31987231
- [Background] Umland EM, Falconieri L. Treatment options for vasomotor symptoms in menopause: focus on desvenlafaxine. Int J Womens Health. 2012;4:305-19. doi: 10.2147/IJWH.S24614. Epub 2012 Jul 5. PMID 22870045
- [Background] Utian WH. Psychosocial and socioeconomic burden of vasomotor symptoms in menopause: a comprehensive review. Health Qual Life Outcomes. 2005 Aug 5;3:47. doi: 10.1186/1477-7525-3-47. PMID 16083502
- [Background] Menopause, 2017, U.S. Food and Drug Administration/Center for Drug Evaluation and Research: Washington, DC. Accessed.